CLINICAL TRIAL: NCT06298955
Title: An Open-Label Study to Evaluate the Long-Term Safety, Tolerability and Efficacy of OMS906 in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Long-Term Safety, Tolerability and Efficacy of OMS906 in Paroxysmal Nocturnal Hemoglobinuria
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS906-PNH-003
Record Dates: First submitted 2024-02-17; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OMS906 study drug (Experimental): OMS906 study drug repeat-dose 5 mg/kg IV administration at 8-week intervals.
  Interventions: Drug: OMS906 study drug

INTERVENTIONS:
Drug: OMS906 study drug — OMS906 study drug repeat-dose 5mg/kg IV administration at 8-week intervals

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of repeat-dose OMS906 5 mg/kg IV administration at 8-week intervals in patients with PNH.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single arm study. The primary objective is to assess the long-term safety and tolerability of OMS906 in patients with PNH. Secondary objectives of this study include assessment of the long-term efficacy of OMS906 in patients with PNH. Patients will receive OMS906 5 mg/kg administered as intravenous (IV) injections at 8-week intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Have completed the last dosing visit of the prior OMS906 PNH study.
2. Female patients of child bearing potential must have a negative result from a highly sensitive urine pregnancy test prior to each dose of OMS906.
3. Females must use highly effective birth control to prevent pregnancy during the clinical trial and for 20 weeks following their last dose of study drug.
4. Males must use highly effective birth control with a female partner to prevent pregnancy during the clinical trial and for 20 weeks after last dose of study drug.
5. Have current vaccination status for Neisseria meningitidis, Streptococcus pneumonia and Hemophilus influenza and agree to maintain vaccination throughout the study.
6. Have provided informed consent

Exclusion Criteria:

1. Platelet count <30,000/µL or absolute neutrophil count <500 cells/µL at the start of the Evaluation Period.
2. Elevation of liver function tests, defined as total bilirubin > 2 x ULN, direct bilirubin > 1.5 x ULN, and elevated transaminases (alanine or aspartate aminotransferase), > 2 X ULN unless due to PNH-related hemolysis.
3. History of any severe hypersensitivity reactions to other monoclonal antibodies or excipients included in the OMS906 preparation.
4. Patients with unresolved serious infections caused by encapsulated bacteria including H. influenzae, S. pneumoniae and N. meningitidis.
5. Pregnant, planning to become pregnant, or nursing female patients.
6. History of any significant medical, neurologic, or psychiatric disorder that in the opinion of the investigator would make the patient unsuitable for participation in the long-term extension.
7. Unable or unwilling to comply with the requirements of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
To assess overall safety and tolerability of OMS906 administration at 8-week intervals in PNH patients. | 104 weeks
  Treatment-emergent adverse events, including clinically significant clinical laboratory tests, 12-lead electrocardiograms, vital signs, and physical examinations recorded as an adverse event.

SECONDARY OUTCOMES:
To assess efficacy measured by hemoglobin (Hgb). | 6 month intervals
  Measured by patients achieving Hb ≥ 12.0 g/dL and by proportion of patients maintaining an increase in Hb ≥ 2 g/dL, achieved in the prior study, through the duration of the long-term extension.
To assess efficacy by transfusion requirements. | Weeks 48 and 96
  Measure proportion of patients who are transfusion free and mean change from baseline in transfusion frequency from the start of the long-term extension.
To assess efficacy by measurement of lactate dehydrogenase (LDH). | Weeks 48 and 96
  Measure mean LDH change from baseline.
To assess efficacy by measurement of reticulocyte count. | Weeks 48 and 96
  Measure mean change in reticulocyte count from baseline.
To assess efficacy by measurement of clinical breakthrough hemolysis. | Weeks 48 and 96
  Measure proportion of patients experiencing clinical breakthrough hemolysis.
To assess population PK Cmax of OMS906. | Weeks 48 and 96
  Pharmacokinetics (PK) of multiple-dose administration of OMS906 using PK parameter maximum concentration (Cmax).
To assess population PK AUC of OMS906. | Weeks 48 and 96
  Pharmacokinetics (PK) of multiple-dose administration of OMS906 using PK parameter area under the time-concentration curve (AUC).
To assess population PK terminal half life of OMS906. | Weeks 48 and 96
  Pharmacokinetics (PK) of multiple-dose administration of OMS906 using terminal half-life parameter.
To assess PD of OMS906 | Weeks 48 and 96
  PD parameters include change from baseline in mature complement factor D (FD).
OMS906 anti-drug antibodies (ADA). | Weeks 24, 48, 72, and 96
  Presence of ADA in serum will be measured.
Assess the change in Functional Assessment of Chronic Illness Therapy (FACIT) fatigue score. | Weeks 24, 48, 72, and 96
  To assess the effect of OMS906 on Quality of Life using the FACIT fatigue scale.

CONTACTS AND LOCATIONS:
Overall Officials: William Pullman, Study Director — Omeros Corporation
Locations (5):
- Germany (2):
  - Omeros Investigational Site, Aachen
  - Omeros Investigational Site, Ulm
- Omeros Investigational Site, Lausanne, Switzerland
- Omeros Investigational Site, Kyiv, Ukraine
- Omeros Investigational Site, Leeds, United Kingdom